CLINICAL TRIAL: NCT05693350
Title: Etiology Of Recurrent Varicose Veins After Stripping Or Ablation Of Superficial
Brief Title: Etiology Of Recurrent Varicose Veins After Stripping Or Ablation Of Superficial Venous System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Tarek Mostafa, Resident Doctor, Assiut University
Other Study IDs: Recurrent Varicose Veins
Record Dates: First submitted 2022-12-02; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Recurrent Varicose Vein of Lower Limb (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DUS — Duplex ultrasound

SUMMARY:
Number of patients and causes and patterns of recurrent varicose veins in the lower limbs in patients with history of varicose veins stripping or ablation of the superficial venous system.

DETAILED DESCRIPTION:
Recurrence of varicose veins following surgery is a common, complex and costly problem in vascular surgery. Despite improvements in preoperative evaluation and methods of treatment, recurrence following varicose vein surgery is reported to occur in between 20 and 80% of cases. Many theories have been put forward concerning the underlying mechanisms and causes. These include poor understanding of the venous anatomy and haemodynamics, inadequate preoperative assessment, inappropriate or incomplete surgery and development of new sites of venous reflux as a consequence of disease progression or neovascularisation. However, it is difficult to evaluate these suggestions since the studies from which they arise vary greatly in their definitions of recurrence, preoperative assessment, initial treatment, classification and method and duration of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1) Ages eligible for the study: 18-60. 2) Sexes eligible for the study: All. 3) Patients with previous intervention for varicose veins. 4) Patients with primary or secondary varicosities. 5) Patient's compliance to follow-up.

Exclusion Criteria:

1) Patients with no history of interventions for varicose veins. 2) Patients treated with injection sclerotherapy alone. 3) Pregnant women. 4) Patients with arterial disease in the same limb (ABI <0.8). 5) Patients with post-thrombotic syndrome

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with previous history of intervention for varicose veins
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Etiology of recurrence of varicose veins in patients previously treated by stripping and ligation or endovenous ablation. | Five years
  Track the recurrence of varicose veins after intervention

SECONDARY OUTCOMES:
Quality of life was assessed by the Aberdeen Varicose Vein Questionnaire (AVVQ) | Five years

REFERENCES:
- [Background] Kostas T, Ioannou CV, Touloupakis E, Daskalaki E, Giannoukas AD, Tsetis D, Katsamouris AN. Recurrent varicose veins after surgery: a new appraisal of a common and complex problem in vascular surgery. Eur J Vasc Endovasc Surg. 2004 Mar;27(3):275-82. doi: 10.1016/j.ejvs.2003.12.006. PMID 14760596
- [Background] Blomgren L, Johansson G, Dahlberg-AKerman A, Noren A, Brundin C, Nordstrom E, Bergqvist D. Recurrent varicose veins: incidence, risk factors and groin anatomy. Eur J Vasc Endovasc Surg. 2004 Mar;27(3):269-74. doi: 10.1016/j.ejvs.2003.12.022. PMID 14760595
- [Background] Hamdan A. Management of varicose veins and venous insufficiency. JAMA. 2012 Dec 26;308(24):2612-21. doi: 10.1001/jama.2012.111352. PMID 23268520